CLINICAL TRIAL: NCT04337996
Title: Dynamic Evaluation of COVID-19 Diagnostic Tests
Acronym: TRODVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RIPH_2020_6
Record Dates: First submitted 2020-04-01; First posted 2020-04-08 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): These are patients whose diagnosis of SARS-Cov-2 infection was made on the Gold-Standard: combined history/clinical examination, PCR and CT scan and requiring hospitalization at Tourcoing Hospital.
  Interventions: Diagnostic Test: COVID-19 diagnostic test

INTERVENTIONS:
Diagnostic Test: COVID-19 diagnostic test — COVID-19 diagnostic tests performed at day 1 (antigen in blood serum, SARS-Cov2 PCR, antibodies in blood serum) COVID-19 diagnostic test performed at day 21 (antibodies in blood serum)

SUMMARY:
Rapid antigenic tests are not yet used in real life. Their contribution in the diagnostic strategy based on the gold standard including anamnesis, thoracic CT and PCR has not been evaluated.

We propose to compare to the Gold-Standard defined above, the combination of an SARS-Cov-2 antigen, anamnesis and thoracic CT for the diagnosis of COVID-19 infection.

DETAILED DESCRIPTION:
This is an interventional study comparing gold standard anamnesis, thoracic CT and PCR versus SARS-Cov-2 antigen, anamnesis and thoracic CT for the diagnosis of COVID-19 infection.

Patients will be sampled for the tests at Day 1 and then monitored for symptoms and clinical data and additional test at Day 21.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patient with confirmed Gold-Standard SARS-CoV-2 (COVID-19) infection
* Presenting at least one criterion for hospitalization:

  * Respiratory failure and oxygenation
  * Circulatory failure (systolic BP < 90 mmHg)
  * Neurological failure (confusion, drowsiness, altered consciousness)
  * Polypathological terrain and co-morbidities (chronic respiratory failure, heart failure or cardiovascular pathology, renal failure, diabetes, immunosuppression, obesity, cirrhosis)
* Eligible for different sampling methods
* Beneficiary of a social insurance scheme or entitled person

Exclusion Criteria:

* Gold Standard not in favour of SARS-Cov-2 infection (COVID 19)
* Minor patient
* Refusal to participate
* Patient under guardianship
* Patient under guardianship
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Comparison of the proportion of patients classified as COVID-19 positive according to the 2 strategies | day 1
  Comparison of the Gold-Standard PCR, anamnesis, thoracic CT scan versus SARS-Cov-2 antigen, anamnesis and thoracic CT scan

SECONDARY OUTCOMES:
Positive or negative Covid-19 test | day 1
  Number of diagnoses invalidated by the antigen + CT scan alone without the contribution of PCR.
Positive or negative character of the antibodies test | day 1
  Comparison of the proportion of patients with positive serology for SARS-Cov2 to the proportion of patients who were classified as COVID-19
Positive or negative character of the antibodies test | day 21
  Comparison of the proportion of patients with positive serology for SARS-Cov2 to the proportion of patients who were classified as COVID-19 at the time of hospitalization
Biological parameters | day 1
  Evolution of biological parameters as a function of time IgM IgA and IgG
Biological parameters | Day 21
  Evolution of biological parameters as a function of time IgM IgA and IgG
medical-economic comparison | day 1
  medical-economic comparison of the first-line use of the antigenic test

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PATOZ, PharmD, Principal Investigator — CH TOURCOING; Barthelemy LAFONDESMURS, MD, Principal Investigator — CH TOURCOING
Locations (1):
- CH Tourcoing, Tourcoing, France

IPD SHARING:
Plan to Share IPD: No